CLINICAL TRIAL: NCT06855628
Title: Assessment Of A Novel Metabolic Imaging Modalities As A Predictor Of Therapeutic Efficacy In Glioblastoma (GBM)
Brief Title: Assessment of Novel Metabolic Imaging Modalities as A Predictor Of Therapeutic EfficacyiIn Glioblastoma (GBM)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-77846; R01CA277832-02 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Glioma; GBM
MeSH Terms: conditions — Glioma | interventions — Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deuterated Glucose + MRI (Experimental): Participants will receive [6,6-²H₂]-glucose orally at a dose of 0.75g per kg of body weight (maximum 60g), dissolved in 200-500mL of water. Approximately 45 minutes after ingestion, participants will undergo an MRI scan consisting of a 30-minute conventional MRI brain study followed by a 1-hour Deuterium Metabolic Imaging (DMI) study. A Gadolinium contrast agent may be administered if more than 4 weeks have passed since the last enhanced MRI scan.
  Interventions: Other: [6,6-²H₂]-Glucose

INTERVENTIONS:
Other: [6,6-²H₂]-Glucose — [6,6-²H₂]-Glucose is a stable isotope-labeled glucose used as a metabolic tracer. It is administered orally to assess glucose metabolism using Deuterium Metabolic Imaging (DMI).
  Other Names: Deuterated Glucose Tracer; Stable Isotope-Labeled Glucose; D-Glucose, [6,6-²H₂]

SUMMARY:
The goal of this study is to evaluate the prognostic capacity of DMI in a trial assessing the efficacy of adding BPM31510, a lipid nano dispersion of CoQ10 to standard treatment of Glioblastoma (GBM).

ELIGIBILITY:
Inclusion Criteria:

* Any participant that consents to entry into the Phase II BPM31510 parent study (BPM31510IV-11)
* Women of childbearing potential must have a negative pregnancy test
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Refuse to have an IV
* Allergy to MRI contrasts
* Diabetic patients who are taking insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 36 months
  Progression-Free Survival (PFS) is defined as the time from the start of treatment until disease progression or death from any cause, whichever occurs first
Overall Survival (OS) | up to 36 months
  Overall Survival (OS) is defined as the time from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lawarence Recht, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States